CLINICAL TRIAL: NCT03468712
Title: Laparoscopic D2 Distal Gastrectomy Following Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancers: A Prospective Multicenter Trial
Brief Title: Laparoscopic D2 Distal Gastrectomy Following Neoadjuvant Chemotherapy for Locally Advanced Gastric Cancers
Acronym: CLASS-03a
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Collaborators: Peking University Cancer Hospital & Institute (Other); Southern Medical University, China (Other); Shanghai Zhongshan Hospital (Other); Chinese PLA General Hospital (Other); Fujian Medical University Union Hospital (Other); Ruijin Hospital (Other); Southwest Hospital, China (Other); RenJi Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Fudan University (Other); Tang-Du Hospital (Other); Harbin Medical University (Other); The First Hospital of Jilin University (Other); Guangdong Provincial People's Hospital (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Jian-Kun Hu, Vice Director of Department of Gastrointestinal Surgery, West China Hospital, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLASS-03a
Record Dates: First submitted 2018-01-23; First posted 2018-03-16 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-03

CONDITIONS: Complications, Postoperative; Surgery--Complications; Cancer of Stomach; Chemotherapy Effect
Keywords: mortality; morbidity; neoadjuvant chemotherapy; laparoscopic gastrectomy; gastric cancer
MeSH Terms: conditions — Postoperative Complications; Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Laparoscopic D2 distal gastrectomy after 3-Cycle XELOX neo-adjuvant chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Laparoscopic D2 distal gastrectomy after 3-Cycle XELOX neo-adjuvant chemotherapy
  Interventions: Procedure: Laparoscopic D2 distal gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic D2 distal gastrectomy — Laparoscopic D2 distal gastrectomy after 3-Cycle XELOX neo-adjuvant chemotherapy

SUMMARY:
Gastric cancer is the third major cancer of global cancer-related death. In China, the early diagnosis rate of gastric cancer is relatively low, and most patients are with locally advanced tumor stage. The neoadjuvant chemotherapy (NAC) can bring the survival advantage for gastric cancer patients with locally advanced tumor stage. The primary goal of NAC is to control the micrometastasis and/or progression of the primary lesion in order to improve potential of radical gastrectomy. NAC is recommended for patients with locally advanced stage (T2-4Nx) according to the latest NCCN Gastric Cancer Guidelines.

Laparoscopy distal gastrectomy (LDG) can achieve a better postoperative short-term recovery than the traditional open distal gastrectomy (ODG), which can reduce the intraoperative blood loss and to shorten the postoperative hospital stay. Therefore, Enhanced Recovery After Surgery program of gastric cancer surgery recommends the use of minimally invasive surgery. For long-term survival outcomes, there is limited evidence supported that laparoscopic gastrectomy is comparable open gastrectomy. Therefore, due to the lack of high-quality prospective clinical trial results, whether advanced tumor is suitable for laparoscopic surgery is still controversial. Therefore, some multi-center prospective randomized controlled trials have been carried out, compared safety and long-term survival outcome between laparoscopic and open gastrectomy in locally advanced gastric cancer patients. CLASS-01 trials reported that for locally advanced gastric cancers, laparoscopic D2 distal gastrectomy is safe and feasible.

Patient's surgical tolerance and stress response may be inhibited after the treatment of NAC. The aim of this trial is to confirm the safety of laparoscopy distal D2 radical gastrectomy for the treatment of after neoadjuvant chemotherapy gastric cancer patients (cT3-4a, N+, M0) in terms of postoperative complications.

DETAILED DESCRIPTION:
This is a prospective, multi-centers, open-label, single-arm study, and the aim of this trial is to evaluate the safety of laparoscopic distal D2 radical gastrectomy for the treatment of locally advanced gastric cancer (cT3-4a, N-/+, M0) after neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* First Round Inclusion Criteria

  1. Age from over 18 to under 75 years;
  2. Primary gastric adenocarcinoma (including pap, tub, muc, sig, and por) confirmed pathologically by endoscopic biopsy;
  3. cT3-4a, N-/+, M0 according to the AJCC 8th Cancer Staging Manual;
  4. Without peritoneal metastasis (examined by laparoscopic examination);
  5. Radical resection (R0) through distal subtotal gastrectomy with D2 lymphadenectomy is anticipated;
  6. Performance status 0 or 1 (Eastern Cooperative Oncology Group) ;
  7. ASA (American Society of Anesthesiology) score ≤ 3;
  8. Normal hemodynamic indices:

  <!-- -->

  1. Blood cell count: HB ≥ 90g/L, ANC ≥ 1.5×109/L, PLT ≥ 80×109/L;
  2. Liver and renal function: BIL<1.5 times of the upper limit of normal reference values, ALT and AST<2.5 times of the upper limit of normal reference values, and Crea≤1 time of upper limits of normal reference values.
* Second Round Inclusion Criteria

  1. Therapeutic response rating after neoadjuvant chemotherapy is CR, PR, SD, or Therapeutic response rating after neoadjuvant chemotherapy is PD, tumor is expected to have radical resection;
  2. Subjects are still willing to continue participating in this clinical trial.

Exclusion Criteria:

* First Round Exclusion Criteria

  1. History of upper abdominal surgery (include endoscopic mucosal resection or endoscopic submucosal dissection, except for laparoscopic cholecystectomy);
  2. History of acute pancreatitis;
  3. Enlarged or bulky regional lymph node (diameter>3cm) by imaging exam;
  4. Patients have received neoadjuvant therapy prior to screen work;
  5. History of other malignant disease within the past five years;
  6. History of cerebrovascular accident within the past six months;
  7. History of continuous systematic administration of corticosteroids within the past month;
  8. Scheduled simultaneous surgery for other disease;
  9. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer;
  10. Pyloric obstruction;
  11. FEV1<50% of predicted value;
  12. Women who are pregnant or lactating at the time of screening;
  13. Severe mental disorder;
  14. Participating in other clinical studies;
  15. Refused to sign the informed consent;
* Second Round Exclusion Criteria

  1. Therapeutic response rating after neoadjuvant chemotherapy is PD, involvement of adjacent structures(T4b), distal metastasis(M1), or enlarged or bulky regional lymph node (diameter>3cm) by preoperative imaging
  2. Patients cannot complete 3 cycles of chemotherapy due to intolerance;
  3. After 3 cycles of neoadjuvant chemotherapy, patients cannot tolerate surgery due to severe adverse reactions, or ASA score ≥ 4 ;
  4. Patients undertake emergency operation due to tumor bleeding, perforation or obstruction during chemotherapy;
  5. After signing the informed consent, the patient withdraws from this clinical trial.

Withdrawal Criteria After Second Round:

1. Intro-abdominal metastasis of primary cancer is revealed intraoperatively;
2. Primary cancer is confirmed to be un-resectable intraoperatively.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2018-03-31 (Actual); Primary Completion 2020-04-30 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative overall morbidity rate | Postoperative 30 days
  The proportion value will be calculated by the number of patients with any operative complication as the numerator and the number of patients undergoing surgical treatment as the denominator.

SECONDARY OUTCOMES:
Postoperative mortality rate | Postoperative 30 days
  Mortality will be calculated as the ratio between the number of patients who died as numerator and number of all patients undergoing surgical treatment as the denominator.
R0 resection rate | The day of surgery
  Number of patients underwent gastrectomy for the denominator, number of R0 resection patients is numerator, the ratio is the R0 resection rate. The definition of R0 resection is according to the Japanese gastric cancer treatment guidelines 2014 (ver. 4)（Gastric Cancer. 2017 Jan;20(1):1-19.）.
Completion rate of laparoscopic surgery | The day of surgery
  Ratio will be calculated with the number of patients complete the laparoscopic gastrectomy as the numerator, and number of all patients undergoing laparoscopic surgical treatment as the denominator.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Kun Hu, M.D. Ph.D., Principal Investigator — West China Hospital
Locations (16):
- China (16):
  - Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Southwest Hospital, the Third Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Harbin Medical University, Harbin, Heilonngjiang
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - RenJi Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai JiaoTong University, Shanghai, Shanghai Municipality
  - Tangdu Hospital, Fourth Military Medical University, Xian, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
Pending

REFERENCES:
- [Background] Hu Y, Huang C, Sun Y, Su X, Cao H, Hu J, Xue Y, Suo J, Tao K, He X, Wei H, Ying M, Hu W, Du X, Chen P, Liu H, Zheng C, Liu F, Yu J, Li Z, Zhao G, Chen X, Wang K, Li P, Xing J, Li G. Morbidity and Mortality of Laparoscopic Versus Open D2 Distal Gastrectomy for Advanced Gastric Cancer: A Randomized Controlled Trial. J Clin Oncol. 2016 Apr 20;34(12):1350-7. doi: 10.1200/JCO.2015.63.7215. Epub 2016 Feb 22. PMID 26903580
- [Background] Schuhmacher C, Gretschel S, Lordick F, Reichardt P, Hohenberger W, Eisenberger CF, Haag C, Mauer ME, Hasan B, Welch J, Ott K, Hoelscher A, Schneider PM, Bechstein W, Wilke H, Lutz MP, Nordlinger B, Van Cutsem E, Siewert JR, Schlag PM. Neoadjuvant chemotherapy compared with surgery alone for locally advanced cancer of the stomach and cardia: European Organisation for Research and Treatment of Cancer randomized trial 40954. J Clin Oncol. 2010 Dec 10;28(35):5210-8. doi: 10.1200/JCO.2009.26.6114. Epub 2010 Nov 8. PMID 21060024
- [Background] Chen XZ, Yang K, Liu J, Chen XL, Hu JK. Neoadjuvant plus adjuvant chemotherapy benefits overall survival of locally advanced gastric cancer. World J Gastroenterol. 2011 Oct 28;17(40):4542-4. doi: 10.3748/wjg.v17.i40.4542. PMID 22110287